CLINICAL TRIAL: NCT07328867
Title: Combined Effects of Dual-task and Perturbation Based Training on Balance and Cognition in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/16
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Balance; Cognition; Fall Risk
Keywords: Physical therapy; Stroke; Perturbation Based Training; Dual-Task Training; Balance; Cognition; Fall risk
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-task and Perturbation Based Training (Experimental): 1. Participants in the experimental group received combined perturbation and dual task training
  2. The intervention was conducted for 3 days a week for 6 consecutive weeks
  3. Each treatment session lasted approximately 40 minutes including 5 minute of warmup and 2 minutes of rest between 2 segments
  4. Primary training modality was treadmill
  5. Initial walking speed was determined individually for each participant by using 10MWT
  6. Perturbations were applied manually during treadmill walking
  7. The intensity of treadmill was progressively increased across sessions by change in directions of perturbations, unpredictability, walking speed and reducing hand support when safe
  8. Dual-task training is added after 3 session and will be performed concurrently with perturbation training.
  9. Cognitive tasks include counting backwards, naming animals, subtracting 3 from 100.
  10. The complexity of the task will progressively increased
  11. Safety should be ensured by using the harness
  Interventions: Procedure: Perturbation + Dual-Task Training
- Perturbation Based Training (Active Comparator): 1. Participants in control group received Perturbation Baesd Training Alone
  2. The intervention was conducted for 3 days a week for 6 consecutive weeks
  3. Each treatment session lasted 40 minutes including 5 minute of warm up and 2 minute of rest between segments
  4. Primary training modality was treadmill
  5. Initial walking speed was determined individually for each participant by using 10MWT
  6. Perturbations were appllied manually during treadmill walking
  7. The intensity of treadmill was progressively increased across sessions by chanfe in directions of perturbations, unpredictability, walking speed and reducing hand support when safe
  8. Safety should be ensured by using the harness, keeping emergency stop at reach, and use of handrails when necessary
  Interventions: Procedure: Perturbation-Based Training

INTERVENTIONS:
Procedure: Perturbation-Based Training — The control group will participate in a structured six-week intervention program consisting exclusively of the Perturbation Based Balance Training. Participants will attend three supervised sessions per week, ensuring consistent oversight and proper technique throughout the program. Each session will began with a warm-up period, followed by two 8-minute segments of perturbation-based treadmill training, with participants allowed a rest period of 60 second to 2 minute between repetitions to prevent fatigue and maintain the quality of each movement. The frequency is maintained consistently, however, perturbations dosage was progressively increased across all six weeks to provide a standardized exposure, allowing for accurate comparison with other intervention groups. Over the entire six-week period, participants will complete a total of 18 supervised sessions, each with three repetitions, summing up to 108 bouts across the intervention.
  Arms: Perturbation Based Training
Procedure: Perturbation + Dual-Task Training — The intervention program spans six weeks and involves both supervised Perturbation sessions and Dual-Task training exercises. Participants will attend three supervised Perturbation based training per week, with each session consisting of two 8-minute segments of the training.
  In addition, participants will perform Dual-Task training and perturbations on treadmill, with each cycle consisting of two segments. This combination of supervised practice will be increased progressively throughout all six weeks. Across the entire program, participants will complete a total of 18 supervised perturbation based balance training and 18 Dual-task training sessions.
  Arms: Dual-task and Perturbation Based Training

SUMMARY:
This study aims to evaluate the Combined Effects of Dual-task and Perturbation Baesd Training on Balance and Cognition in Stroke Patients. Stroke is an acute cerebrovascular disorder that can impair cognitive, motor, and balanace abilites. Stroke is the second largest cause of death and disability globally. According tp studies, people who have had a stroke are more likely to fall than others who are same age and gender. PBBT is known as artificially induced balance training technique that can mimics the loss of balance that can occur naturally in freal life. Reduction in falls has been reported broadly by the use of perturbation based balance training. Current study will be and RCT on 33 participants based on the inclusion critieria. Participants will be randomly and equally divided into two groups; group B receiving Perturbation Based Training Alone and Group A receiving Dual-task and Perturbation Based Balance Training. The treatment will be given for 40 minutes, 3 days a week for 6 consecutive weeks. The assessment will be conducted at baseline, for cognition by Montreal Cognitive Assessment Scale (MoCA), for initial treadmill speed 10 Meter Walk Test (10MWT), for balance by Berg Balance Scale (BBS), and for fall riak by Fall Efficacy Scale (FES). Final assessment will be conducted after 6 weeks.

DETAILED DESCRIPTION:
Stroke is a multifaceted disease that can be caused by a variety of risk factors, disease processes and causes. Stroke results in the change of cognitive function, which effects resulting in minor impairment to the development of post-stroke dementia. The cognitive deficiencies in a stroke survivors have significant influence on their daily productivity. In addition, falls are a prevalent and potentially fatal issue for as many as 47% of all stroke patients admitted to the hospital.Some studies suggest that Dual-task training when paired with mechanical action of treadmill could maximize the constraint on the cognitive control processes for gait.

ELIGIBILITY:
Inclusion Criteria:

* No limitation of genders.
* Age between 25-80 years
* Participants diagnosed with chronic stroke
* Participants being able to walk with or without walking aid independently or under supervision
* Participants with impaired balance as indicated by a score of <=41 on BBS
* Participants with Montreal Cognitive Assessment Score <26

Exclusion Criteria:

* Patient with sinificant co morbidties or secondary complications including orthopedic or rheumatological disorders were excluded
* Patients with severe cognitive impairment or dementia
* Apraxia or hemi-neglect
* Participants with body weight >100kg
* Participants with significant visual or hearing impairments
* Patients with epilepsy or pacemaker
* Participants with peripheral or central neuropathies that could impair balance

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2025-06-14 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Balance | 6 weeks
  Berg Balance Scale (BBS) was used, Maximum Total=56 points (41-56=Low fall risk, 21-40= Medium fall risk, 0-20 High fall risk)
Cognition | 6 weeks
  Montreal Cognitive Assessment Scale, Maximum score=30 (26-30= normal cognition, 18-25= mild cognitive impairment, 10-17 moderate cognitive Impairment, <10=severe cognitive impairment

SECONDARY OUTCOMES:
Fall Risk | 6 Weeks
  Fall Efficacy Scale (FES), Total score=10-100 (higher score = greater fear of falling

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan